CLINICAL TRIAL: NCT00880854
Title: Phase I Dose-escalation Trial of CP-675,206 (Tremelimumab, Anti-CTLA-4 Monoclonal Antibody) for Patients With BCG-resistant Localized Transitional Cell Carcinoma of the Bladder
Brief Title: Study of CP-675,206 in Bacillus Calmette-Guerin (BCG)-Resistant Bladder Cancer
Status: Withdrawn | Phase: Phase 1 | Type: Interventional
Why Stopped: Lack of accrual
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CO08807; NCI-2011-03676 (Registry Identifier: NCI Trial ID); H-2008-0227 (Other: Institutional Review Board); A534260 (Other: UW Madison); SMPH/MEDICINE/MEDICINE*H (Other: UW Madison)
Record Dates: First submitted 2009-04-13; First posted 2009-04-14 (Estimated); Last update posted 2019-11-15 (Actual); Status verified 2019-11

CONDITIONS: Bladder Cancer
Keywords: bladder cancer; BCG-resistant localized transitional cell of the bladder
MeSH Terms: conditions — Urinary Bladder Neoplasms | interventions — tremelimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- 1 (Experimental): BCG 81 mg intravesical weekly x 6 beginning on week 1, and weekly x 3 beginning at week 15 in combination with CP-675,206 I.V. week 3, week 1
  Interventions: Drug: BCG and CP-675,206

INTERVENTIONS:
Drug: BCG and CP-675,206 — Dose level -1: BCG 81 mg intravesical weekly x 6 beginning on week 1, and weekly x 3 beginning at week 15 CP-675,206 3 mg/kg I.V. week 3, week 15
  Dose level 1: BCG 81 mg intravesical weekly x 6 beginning on week 1, and weekly x 3 beginning at week 15 CP-675,206 6 mg/kg I.V. week 3, week 15
  Dose level 2: BCG 81 mg intravesical weekly x 6 beginning on week 1, and weekly x 3 beginning at week 15 CP-675,206 10 mg/kg IV week 3, week 15
  Dose level 3: BCG 81 mg intravesical weekly x 6 beginning on week 1, and weekly x 3 beginning at week 15 CP-675,206 15 mg/kg IV week 3, week 15
  Other Names: Bacille Calmette-Guerin (BCG); Tremelimumab

SUMMARY:
The purpose of this study is to find out the highest safe dose of the investigational drug CP-675,206 when given in combination with BCG therapy to patients who have experienced recurrent superficial bladder cancer after standard BCG treatment.

In addition, the study will look to see if taking CP 675,206 generates an immune response and evaluate how the drug affects superficial bladder cancer.

ELIGIBILITY:
Inclusion Criteria:

* Histologic diagnosis of transitional cell cancer of the bladder must have completed a transurethral resection of all visible bladder tumors, and have completed two previous 6-week courses with intravesical BCG.
* Evidence of disease recurrence within 1 year of previous BCG treatment
* Tumor tissue must be available from biopsy for study related immunohistochemical analysis
* If sexually active must use reliable form of contraception while on study and for 4 weeks after last treatment
* ECOG performance status of <2
* Life expectancy of at least 6 months
* Adequate hematologic, renal and liver function
* Informed consent

Exclusion Criteria:

* No evidence of immunosuppression or treated with immunosuppressive therapy within 6 months
* No prior radiation to the pelvis
* No gross hematuria within 1 week prior to planned week 1 treatment
* Cannot have previous intolerance to BCG
* Cannot be seropositive for HIV, hepatitis B(HBV) or hepatitis C(HCV) per patient history
* No evidence of metastatic disease
* No prior treatment with anti-CTLA-4 monoclonal antibody
* Can not be pregnant or lactating
* No history of autoimmune disorder
* No history of thyroid or adrenal insufficiency
* No history of inflammatory bowel conditions, including diverticulitis, ulcerative colitis, Crohn's or celiac disease, intractable urinary tract infection

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2009-06; Primary Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
To determine the safety of CP-675,206 when delivered in combination with BCG in patients with BCG-resistant bladder carcinoma in situ | 24 months

SECONDARY OUTCOMES:
To determine whether patients treated with CP-675,206 in combination with BCG develop cancer antigen-specific systemic immune responses | 24 months
To determine whether patients treated with CP-675,206 in combination with BCG develop an increase in tumor-infiltrating lymphocytes | 24 months
To determine whether patients treated with CP-675,206 in combination with BCG develop pathological and cytological complete responses | 24 months
To determine the 1-year recurrence-free survival | 24 months
To determine a recommended dose and schedule for phase II trial evaluation based on the maximum tolerated dose | 24 months

CONTACTS AND LOCATIONS:
Overall Officials: Douglas G McNeel, M.D., Ph.D., Principal Investigator — University of Wisconsin, Madison

REFERENCES:
- See also: University of Wisconsin Carbone Cancer Center — https://cancer.wisc.edu/